CLINICAL TRIAL: NCT06987487
Title: Implementazione Della Job Rotation Per lo Sviluppo Delle Competenze Infermieristiche e il Miglioramento Della Salute Organizzativa in un Dipartimento di Scienze Cardiovascolari: Un Protocollo di Ricerca
Brief Title: Implementation of Job Rotation for the Development of Nursing Competencies and the Improvement of Organizational Health in a Department of Cardiovascular Sciences: A Research Protocol
Acronym: JR_01
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Manuela Cavalletti, Nursing Director, Principal Investigator, Dr., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ID7538; Prot. 0000612/25 (Other: Fondazione Policlinico Universitario A. Gemelli IRCCS)
Record Dates: First submitted 2025-05-09; First posted 2025-05-23 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Job rotation; Professional competence; Clinical competence; Job satisfaction; Burnout; Organizational health; Cardiovascular nursing
MeSH Terms: conditions — Burnout, Psychological | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: A two-arm, non-randomized, parallel assignment study comparing nurses participating in a structured job rotation program with nurses continuing standard work routines within a cardiovascular department.
Masking Description: Due to the nature of the organizational intervention, neither participants nor investigators are blinded to group assignment. Nurses are aware of their participation in the job rotation program, and data collection is conducted openly by the research team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Job Rotation Group (Experimental): Nurses in this group will participate in a structured job rotation program involving bimonthly rotations across various units in the Department of Cardiovascular Sciences, including intensive care, medical, surgical, and rehabilitation units. The intervention aims to enhance clinical and professional competencies, organizational health, and reduce burnout.
  Interventions: Behavioral: Job Rotation Program
- No Job Rotation (Other): Nurses in this group will continue performing their usual clinical duties in their original units, without participating in the job rotation program. This group will be used as a comparator to assess the effects of the intervention.
  Interventions: Behavioral: No Job Rotation (Standard Care)

INTERVENTIONS:
Behavioral: Job Rotation Program — Nurses assigned to the intervention group will participate in a structured job rotation program across multiple cardiovascular units (e.g., intensive care, medical, surgical, rehabilitation) every two months for a period of 12 months. Each rotation cycle involves temporary reassignment to a different unit, followed by a return to the original unit. Each nurse will undergo orientation and receive support from a dedicated tutor in the host unit.
  Arms: Job Rotation Group
Behavioral: No Job Rotation (Standard Care) — Nurses in the control group will continue their usual duties in their respective units without participating in the job rotation program. They will be exposed to the same data collection tools as the intervention group, but without any planned rotation or inter-unit movement.
  Arms: No Job Rotation

SUMMARY:
This prospective, monocentric observational study aims to evaluate the implementation of a Job Rotation (JR) program in the Department of Cardiovascular Sciences at Fondazione Policlinico Universitario A. Gemelli IRCCS. The primary objective is to assess the impact of JR on the development of professional and clinical nursing competencies, as well as on organizational health and burnout levels. The study involves two groups of nurses: one participating in a structured JR program with bimonthly rotations across intensive, medical, surgical, and rehabilitation units; and a control group continuing routine activities. Outcomes will be measured using validated tools, including the Italian Nurse Competence Scale - Short Form (I-NPCS-SF), the Italian Nurse Competence Scale (INCS), the Maslach Burnout Inventory - HSS, and the QISO questionnaire. The research investigates whether JR improves competency, reduces burnout, and enhances perceived organizational health.

DETAILED DESCRIPTION:
Job Rotation (JR) is an organizational practice where employees are periodically transferred between roles, departments, or different tasks within the same organization. This approach has been adopted in various sectors to promote flexibility, foster the development of new skills, and maintain existing competencies. It also helps reduce job monotony and enhances professional engagement. In the healthcare field, particularly in nursing, JR is emerging as a promising strategy to address key challenges such as burnout, staff shortages, and the need to adapt quickly to dynamic and complex care environments.

In specialized areas such as cardiology, which includes intensive care, medical-surgical units, and cardiac rehabilitation, JR can support the development of transversal competencies in emergency management, the use of advanced technologies, and interprofessional collaboration. The alternating roles allow nurses to gain practical skills and a comprehensive understanding of the patient care pathway, ultimately improving care quality and emergency responsiveness.

Implementing a JR protocol in a Department of Cardiovascular Sciences may foster a more flexible and competent nursing workforce and promote a collaborative and resilient work environment. Periodic transfers between specialized areas may help nurses broaden their competencies, better adapt to workload variations, and improve both operational efficiency and job satisfaction. JR could also enhance team cohesion and mutual support, reducing long-term adverse events and improving care quality.

Primary Objective To assess the impact of Job Rotation (JR) in the Department of Cardiovascular Sciences on nursing professional and clinical competencies, organizational health, and burnout levels.

Secondary Objectives To evaluate the effectiveness of JR in maintaining or improving professional and clinical nursing competencies.

To measure differences in mean competency scores between JR and non-JR nurses. To analyze the relationship between the number of JR cycles completed and competency levels.

To assess the impact of JR on organizational health and nurse burnout.

Primary Endpoint Difference in professional and clinical competency levels across specialized units (cardiac intensive care, cardiac surgery ICU, medical, surgical, and cardiac rehabilitation units) between JR and non-JR groups, using the Italian Nurse Competence Scale - Short Form (I-NPCS-SF).

Secondary Endpoints Mean job satisfaction score among nurses. Differences in burnout levels (Maslach Burnout Inventory - Human Services Survey) between JR and non-JR groups.

Differences in perceived organizational health (QISO) between JR and non-JR groups.

Relationship between the number of JR cycles and clinical competency scores.

Hypotheses H1: JR improves professional and clinical nursing competencies. H2: JR nurses achieve higher competency scores than non-JR nurses. H3: Nurses completing more JR cycles show greater competency improvement. H4: JR enhances organizational health. H5: JR reduces nurse burnout.

Methods

Design:

Prospective, single-center, observational study without drugs or medical devices.

Duration: 12 months from ethics approval and administrative clearance until data saturation.

Setting: Fondazione Policlinico Universitario A. Gemelli IRCCS - Department of Cardiovascular Sciences.

This study will involve the following units:

Cardiovascular Rehabilitation (7M) Coronary Intensive Care Unit (8C) Cardiac Anesthesia and Intensive Care (8N) Cardiology and Electrophysiology (8L) Internal Cardiovascular Medicine and Heart Failure (8M) Cardiac Surgery (8P) Vascular Surgery and Cardiology (9L)

Conceptual Framework Based on the preliminary literature review, JR appears to have a positive impact on the development of clinical nursing competencies, improving job satisfaction and organizational health while reducing perceived burnout. The conceptual model illustrates the relationships among study variables.

Intervention The JR program involves bimonthly rotations. One nurse from each unit will be transferred to another participating unit. At the end of each cycle, the nurse returns to their original unit, and a new nurse begins rotation. This cyclic mechanism continues throughout the study duration.

Training needs will be identified by the Principal Investigator with support from unit coordinators. A tutor may be assigned if needed. Training will follow the hospital's standard operational instruction for onboarding.

Data Collection Procedure Pre-intervention: All tools will be administered to both intervention and control groups.

Post-intervention: Final assessment will be administered to the intervention group to evaluate changes in competencies, satisfaction, burnout, and organizational health.

Sample Size and Statistical Analysis Sample size was calculated using G*Power with a significance level of 0.05, power of 0.9, and effect size of 0.5, resulting in a required sample of 86 participants (43 per group).

Data analysis will include:

Descriptive statistics: frequencies, percentages, means ± SDs or medians with IQRs.

Normality testing using skewness, kurtosis, and Shapiro-Wilk test. Between-group comparisons: Student's t-test (for normal data), Mann-Whitney U test (for non-normal data), chi-square or Fisher's exact test (for categorical data).

Within-group comparisons (JR group pre/post): paired t-test or Wilcoxon test. Repeated measures analysis: ANOVA or Kruskal-Wallis test, depending on distribution.

Correlation analysis: Pearson or Spearman, based on data distribution. Significance threshold set at p < 0.05. Analyses will be conducted using SPSS and R.

Safety and Adverse Event Management The JR program will be structured to ensure nurse and patient safety during transitions. Pre-rotation training will cover safety protocols, technologies, and emergency procedures. A peer tutor will support each nurse during initial integration. Continuous monitoring of safety and performance will be conducted. Adverse events will be reported through the hospital's incident reporting system, and corrective actions will be taken as needed.

Expected Results JR is expected to enhance nurses' clinical and professional competencies, reduce burnout, and improve organizational health and job satisfaction. By fostering cross-unit collaboration, JR may also contribute to greater cohesion, lower absenteeism, and better workload management. The intervention may support a more adaptable and efficient workforce, ultimately improving care quality and clinical outcomes.

Coercion and Undue Influence Risk Mitigation The study complies with internal policies to safeguard employee rights, including informed decision-making and freedom from coercion or negative professional consequences. Adequate time and support will be given to participants before consent is obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Registered nurses employed in the Department of Cardiovascular Sciences at Fondazione Policlinico Universitario A. Gemelli IRCCS
2. Willing and able to provide written informed consent
3. Willing to participate in the job rotation program or remain in their original unit, depending on group assignment

Exclusion Criteria:

1. Nurses with certified physical or psychological limitations that prevent participation in job rotation
2. Nurses who do not provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Change in clinical and professional nursing competence | JR group: T0 (baseline) and T1 (2 months, end of rotation); Control group: T0 only (baseline)
  Competence will be assessed using the Italian Nurse Competence Scale - Short Form (I-NPCS-SF). All participants (JR and control groups) will complete the assessment at baseline (T0). Only the Job Rotation (JR) group will complete a second assessment after the rotation period (T1, 2 months). The higher the overall I-NPCS-SF score (%), the higher the clinical and/or professional competencies.

SECONDARY OUTCOMES:
Change in job satisfaction | JR group: T0 (baseline) and T1 (2 months, end of rotation); Control group: T0 only (baseline)
  Job satisfaction will be assessed using the QISO questionnaire (Nursing Questionnaire on Organizational Health), which specifically addresses this construct. The measure will be collected at baseline (T0) in both groups and at T1 (2 months) in the JR group only.
  The questionnaire consists of 118 items designed to explore 14 theoretical dimensions of organizational well-being and three groups of indicators (positive, negative, and psychophysical distress) within the nursing population. Except for the first and last sections-dedicated to collecting sociodemographic data and open-ended responses-the items use a 4-point Likert scale ranging from "never"/"insufficient" (score 1) to "often"/"good" (score 4). Higher scores indicate better organizational health. A cutoff score of 2.6 is used to assess overall organizational well-being and to determine the presence or absence of specific workplace phenomena across the different dimensions.
Change in burnout levels | JR group: T0 (baseline) and T1 (2 months, end of rotation); Control group: T0 only (baseline)
  Burnout will be measured using the Maslach Burnout Inventory (MBI) - Human Services Survey (HSS). Both groups will be assessed at T0; only the JR group will be reassessed at T1.
  The MBI-HSS yields three distinct scores, each corresponding to a core dimension of burnout: Emotional Exhaustion (EE), Depersonalization (DP), and Personal Accomplishment (PA). High levels of burnout are typically indicated by elevated scores in EE and DP combined with a low score in PA. Each score is interpreted based on its position within the normative distribution: values in the upper third are classified as high, those in the middle third as moderate, and those in the lower third as low.
Change in perceived organizational health | JR group: T0 (baseline) and T1 (2 months, end of rotation); Control group: T0 only (baseline)
  Organizational health will be measured using the QISO questionnaire (Nursing Questionnaire on Organizational Health), which specifically addresses this construct. All participants will be assessed at T0 (baseline); only the JR group at T1 (after 2 months).
  The questionnaire consists of 118 items designed to explore 14 theoretical dimensions of organizational well-being and three groups of indicators (positive, negative, and psychophysical distress) within the nursing population. Except for the first and last sections-dedicated to collecting sociodemographic data and open-ended responses-the items use a 4-point Likert scale ranging from "never"/"insufficient" (score 1) to "often"/"good" (score 4). Higher scores indicate better organizational health. A cutoff score of 2.6 is used to assess overall organizational well-being and to determine the presence or absence of specific workplace phenomena across the different dimensions.
Association between number of completed rotation cycles and competence scores (JR group only) | Baseline (prior to the first rotation cycle) and at the end of each subsequent bimonthly cycle, if applicable.
  The number of completed job rotation cycles-treated as a continuous independent variable-will be analyzed to assess its association with clinical and professional competence scores. Each nurse may complete more than one rotation during the intervention period. Competence will be measured at the end of each cycle.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the nature of the study involving healthcare professionals as participants. Although data will be pseudonymized, the limited sample size and organizational setting may pose a risk of indirect re-identification. Additionally, the informed consent did not include provisions for data sharing outside the research team.

REFERENCES:
- [Background] Platis C, Ilonidou C, Stergiannis P, Ganas A, Intas G. The Job Rotation of Nursing Staff and Its Effects on Nurses' Satisfaction and Occupational Engagement. Adv Exp Med Biol. 2021;1337:159-168. doi: 10.1007/978-3-030-78771-4_18. PMID 34972902
- [Background] Liang HY, Tang FI, Wang TF, Yu S. Evaluation of Nurse Practitioners' Professional Competence and Comparison of Assessments Using Multiple Methods: Self-Assessment, Peer Assessment, and Supervisor Assessment. Asian Nurs Res (Korean Soc Nurs Sci). 2021 Feb;15(1):30-36. doi: 10.1016/j.anr.2020.10.004. Epub 2020 Nov 26. PMID 33249140
- [Background] Kim HY. Statistical notes for clinical researchers: assessing normal distribution (2) using skewness and kurtosis. Restor Dent Endod. 2013 Feb;38(1):52-4. doi: 10.5395/rde.2013.38.1.52. Epub 2013 Feb 26. No abstract available. PMID 23495371
- [Background] Ho WH, Chang CS, Shih YL, Liang RD. Effects of job rotation and role stress among nurses on job satisfaction and organizational commitment. BMC Health Serv Res. 2009 Jan 12;9:8. doi: 10.1186/1472-6963-9-8. PMID 19138390
- [Background] Emanuela P, Alessandro S, Florian S, Gennaro R, Ina D, Rosario C, Ippolito N. Psychometric Validation of the Nursing Professional Competence Scale Among Italian Nurses and Albanian Nursing Students. J Nurs Meas. 2023 Nov 29;31(4):595-605. doi: 10.1891/JNM-2021-0060. PMID 37558253
- [Background] Chatterjee S, Shah A, Sharma R, Wadhwa M. Effect of Job Rotation Concept for Nursing Staff with Special Reference to Private Based Hospital, Vadodara. Indian J Occup Environ Med. 2023 Jul-Sep;27(3):197-204. doi: 10.4103/ijoem.ijoem_354_21. Epub 2023 Oct 6. PMID 38047175
- [Background] Celikturk Doruker N, Demir Korkmaz F. Investigation of burnout and quality of work life of cardiac surgery nurses: A cross-sectional study. Nurs Crit Care. 2024 Nov;29(6):1373-1384. doi: 10.1111/nicc.13124. Epub 2024 Jul 14. PMID 39004602
- [Background] Ioannou P, Katsikavali V, Galanis P, Velonakis E, Papadatou D, Sourtzi P. Impact of Job Satisfaction on Greek Nurses' Health-Related Quality of Life. Saf Health Work. 2015 Dec;6(4):324-8. doi: 10.1016/j.shaw.2015.07.010. Epub 2015 Aug 20. PMID 26929845
- [Background] Bagnasco A, Barisone M, Aleo G, Watson R, Catania G, Zanini M, Thompson DR, Sasso L. An international e-Delphi study to identify core competencies for Italian cardiac nurses. Eur J Cardiovasc Nurs. 2021 Oct 27;20(7):684-691. doi: 10.1093/eurjcn/zvab003. PMID 33595064
- [Background] Alfuqaha OA, Al-Hairy SS, Al-Hemsi HA, Sabbah AA, Faraj KN, Assaf EM. Job rotation approach in nursing profession. Scand J Caring Sci. 2021 Jun;35(2):659-667. doi: 10.1111/scs.12947. Epub 2020 Dec 16. PMID 33326130
- [Background] Alexandrou M, Simsek B, Rempakos A, Kostantinis S, Karacsonyi J, Rangan BV, Mastrodemos OC, Allana SS, Rao SV, Linzer M, Egred M, Milkas A, Sandoval Y, Burke MN, Brilakis ES. Burnout in cardiology: a narrative review. J Invasive Cardiol. 2024 May;36(5). doi: 10.25270/jic/23.00292. PMID 38422526
- See also: Maslach burnout inventory instruments and scoring guides forms. http://www.mindgarden.com — http://www.mindgarden.com